CLINICAL TRIAL: NCT05878730
Title: A Case-control Study Comparing Melatonin Nocturnal Secretion Between Lithium Responders Versus Non Responders in Type 1 Bipolar Disorder.
Brief Title: Melatonin and Response to Lithium
Acronym: MeLiR
Status: Recruiting | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: APHP221168; 2022-A02550-43 (Other: ID RCB Number)
Record Dates: First submitted 2023-05-19; First posted 2023-05-26 (Actual); Last update posted 2025-08-08 (Actual); Status verified 2025-08

CONDITIONS: Bipolar Disorder I
Keywords: lithium
MeSH Terms: interventions — Urine Specimen Collection

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- good-responders (GR) to lithium in euthymic BD-1 individuals
  Interventions: Diagnostic Test: urine collection; Diagnostic Test: Level of Proteins; Diagnostic Test: Level of mRNA and miRNA; Diagnostic Test: Level of plasmatic and intraerythrocytic lithium
- non-responders (NR) to lithium in euthymic BD-1 individuals
  Interventions: Diagnostic Test: urine collection; Diagnostic Test: Level of Proteins; Diagnostic Test: Level of mRNA and miRNA; Diagnostic Test: Level of plasmatic and intraerythrocytic lithium

INTERVENTIONS:
Diagnostic Test: urine collection — * Urine collection will be made on a 12 hours period (20h00-8h00), the night before V2
  * at V2 : 2 mL urinal sample for measure of 6-SMT concentration (ng/mL) and creatinin (mg/mL)
  * Measure of 6-SMT will be made by a validated radio-immunology assay
Diagnostic Test: Level of Proteins — * blood sample at V2 (2x3.5mL citrate tubes)
  * measured by ELISA
Diagnostic Test: Level of mRNA and miRNA — * blood sample at V2 (2x2.5mL PAX-gene tube)
  * measured by quantitative RT-PCR
Diagnostic Test: Level of plasmatic and intraerythrocytic lithium — * blood sample at V2 (mmol/L)
  * 4mL EDTA tube

SUMMARY:
Bipolar disorders are mental illnesses characterized by the recurrence of mood-episodes, that can have a severe impact on the life of individuals. The effect of lithium, one of the main medications used to treat acute episodes or prevent them from happening, is very different from one individual to an-other. So far, there is no way to predict in advance for whom patient this treatment will be effective or for whom it will not.

Finding markers that can predict as early as possible the efficiency of this treatment is a major field of current research in psychiatry, in order to avoid maintaining an inefficient treatment for several years that can have negative side-effects.

Over the past decades, it has been shown by multiple studies that lithium can act on the biological clock, that regulates circadian rhythmicity of the body (i.e. rhythms that presents a 24 hours periods, such as rhythms of sleep and activity, feeding, social activities...). But it is still very unclear whether the effect of lithium in regulating the mood in bipolar disorders is mediated by this action.

Melatonin is one of the key-regulator of circadian rhythmicity of the human body. Our hypothesis, based on some previous studies, is that the action of lithium in type-1 bipolar disorder (BD-I) is related to an action on melatonin secretion.

To test that, we want in this study to compare the noctunal secretion of melatonin between BD-I individuals with a good response to lithium versus with a poor response to lithium.

DETAILED DESCRIPTION:
The study is a monocentric case-control study comparing the level of urinary nocturnal secretion of 6-sulfatoxy-melatonin between good-responders (GR) and non-responders (NR) to lithium in euthymic BD-1 individuals.

The study will also compare the levels of 14-3-3 proteins and miR-451 between these two groups. They are regulators of melatonin-synthesis, that on one hand have been previously associated in autism spectrum disorders to melatonin level modifications and on the other hand have been shown in one preclinical study in rat to be regulated by a lithium treatment.The study also compare the levels of other proteins and mRNA of interest related to ciracdian regulatory pathways.

Euthymic BD-1 patients treated by lithium will be pre-selected and lithium response will be assessed by clinicians using the validated ALDA-scale.

V1 = inclusion (D0) :

* assessment of inclusion and exclusion criteria
* written consent
* collection of socio-demographic data, clinical data
* questionaries : MADRS (Montgomery-Absberg Depressive scale for depressive symptoms), YMRS (Young Mania Rating Scale for manic symptoms), Berlin score (risk of undiagnosed obstructive sleep apnea)
* ALDA scale for assessment of lithium response
* information and furniture for one-night urine collection and one-week sleep diary
* planning of V2, the day after diurnal urine collection

V2 (D8 to D30):

* collection of the urine collection and the sleep diary
* blood sample for measure of plasmatic level of lithium, 14.3.3 proteins and miR-451, mRNA or proteins of interest
* Self-questionaries : PSQI (Pittsburg Sleep Quality Index for sleep assesment), CSM (Composite Scale of Morningness for assessment of morning vs evening chronotype), CTI (Circadian Type Inventory for assessment of chronotype)

ELIGIBILITY:
Inclusion Criteria:

* BD-1 as defined by DSM-5
* Age : 18 to 70
* Current treatment by lithium for more than one year
* Euthymia defined by : MADRS <8 and YMRS <8 at inclusion ; no hospitalization or change in mood-stabilizing treatment in the previous 3 months
* Health condition compatible with blood and urinal sampling
* Being affiliated to french social security
* Written consent

Exclusion Criteria:

* Treatment by : melatonin, agomelatin, benzodiazepines or hypnotic in the last 15 days
* Treatment by a strong CYP1A2 inducer in the last month : ciprofloxacine, dihydralazine, fluvoxamine, norfloxacine
* Current substance use disorder except for tobacco
* Chronic renal failure with glomerular filtration rate <60mL/min
* Jetlag in the last 15 days or life-event impacting circadian rhythmicity (birth, grief, night-work...)
* Sleep disorders such as Obstructive Sleep-Apnea, restless leg syndrome, narcolepsy
* Pregnancy, breastfeeding
* Guardianship
* Inability to understand french, illiteracy

Ages: 18 Years to 70 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Euthymic BD-1 patients treated by lithium
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2023-07-26 (Actual); Primary Completion 2026-07 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Ratio between 6-sulfatoxy-melatonin (6-SMT) concentration and creatinin concentration on a 12-hours nocturnal urine collection | at day 30
  Ratio between 6-sulfatoxy-melatonin (6-SMT) concentration and creatinin concentration on a 12-hours nocturnal urine collection (8pm to 8am) :
  * Urine collection will be made on a 12 hours period (20h00-8h00), the night before D30
  * at D30 : 2 mL urinal sample for measure of 6-SMT concentration (ng/mL) and creatinin (mg/mL)
  * Measure of 6-SMT will be made by a validated radio-immunology assay

SECONDARY OUTCOMES:
Level of Proteins | at day 30
  Level of Proteins (including protein 14.3.3) in ng/mL :
  * blood sample at D30 (2x3.5mL citrate tubes)
  * measured by ELISA
Level of mRNA and miRNA | at day 30
  Level of mRNA and miRNA (including miR-451)
  * blood sample at D30 (2x2.5mL PAX-gene tube)
  * measured by quantitative RT-PCR
Level of plasmatic and intraerythrocytic lithium | at day 30
  Level of plasmatic and intraerythrocytic lithium (mmol/L)
  * blood sample at D30 (mmol/L)
  * 4mL EDTA tube

CONTACTS AND LOCATIONS:
Locations (1):
- Hôpital Fernand-Widal, Paris, Île-de-France Region, France

IPD SHARING:
Plan to Share IPD: No